CLINICAL TRIAL: NCT02189590
Title: A Randomized Comparison of the I-gel and Air-Q as Conduits for Fiberoptic-guided Tracheal Intubation in Children
Brief Title: Assessment of the I-gel and Air-Q Supraglottic Airways as Conduits for Tracheal Intubation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Narasimhan Jagannathan, Primary Investigator; MD, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: I-gel versus air-Q
Record Dates: First submitted 2014-07-09; First posted 2014-07-14 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Tracheal Intubation in Children
Keywords: supraglottic airway; children; fiberoptic guided tracheal intubation; air-Q; i-gel

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- air-Q (Experimental): Patients will receive the air-Q with size based on manufacturer recommendations of body weight
  Interventions: Device: air-Q
- i-gel (Experimental): Patients will receive the i-gel with size based on manufacturer recommendations of body weight
  Interventions: Device: i-gel

INTERVENTIONS:
Device: i-gel — Patients randomized to this intervention will have the i-gel placed following induction of general anesthesia. Subsequent tracheal intubation will be performed using the device as a conduit for fiberoptic-guided intubation. Following successful tracheal intubation, the device will be removed.
  Arms: i-gel
Device: air-Q — Patients randomized to this intervention will have the air-Q placed following induction of general anesthesia. Subsequent tracheal intubation will be performed using the device as a conduit for fiberoptic-guided intubation. Following successful tracheal intubation, the device will be removed.
  Arms: air-Q

SUMMARY:
The purpose of this study is to determine if there is a difference in time for successful fiberoptic guided tracheal intubation through the i-gel or air-Q supraglottic airway.

DETAILED DESCRIPTION:
The goal of this randomized study is to evaluate the efficacy of the i-gel as a conduit for fiberoptic tracheal intubation when compared to the air-Q in children. Intubations will be performed by residents in training. The primary outcome is of time for successful tracheal intubation. The investigators hypothesize that residents will intubate the trachea faster when using the air-Q as compared to the i-gel. The ease of placement of the supraglottic airway device, fiberoptic grade of laryngeal view, time for device removal after intubation, and peri-operative complications will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing general anesthesia requiring tracheal intubation
* Age one month to six years

Exclusion Criteria:

* ASA class IV, V
* Children receiving emergent surgery
* History or high suspicion of a difficult airway
* Active upper respiratory tract infection

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Time to Successful Tracheal Intubation | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Time to successful tracheal intubation when using fiberoptic bronchoscopy to intubate through the i-gel or air-Q ILA. Three separate times will be measured by an independent observer: 1) Time to first glottic view: defined as the duration of time ending with the first view of the glottic opening. 2) Time to carinal view: defined as the duration of time ending with visualization of the carina. 3) Time to successful tracheal intubation: defined as the duration of time ending with the observation of a square wave end-tidal capnogram after successful tracheal intubation

SECONDARY OUTCOMES:
Ease of Placement of Supraglottic Airway | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Ease of placement of supraglottic device ranging from 1 (easy) to 4 (difficult).
Number of Attempts to Place the Supraglottic Device | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Number of attempts will be limited to 3
Supraglottic Airway Leak Pressure | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The airway pressure at which an airway leak is observed after placement of the supraglottic airway
Fiberoptic Grade of Laryngeal View | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Fiberoptic Grade of Laryngeal View through either the air Q or i-gel will be graded using a previously published grading system
Airway Maneuvers | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  The number and type of airway maneuvers performed during tracheal intubation will be recorded
Postoperative Complications | Participants will be followed for the duration of anesthesia and 24 hours postoperatively
  Complications noted postoperatively relating to the airway, such as sore throat or hoarseness.
Time to Placement of Supraglottic Airway | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Time to placement of supraglottic device will be measured.
Number of Attempts to Place the Tracheal Tube | participants will be followed for the duration of anesthesia and after surgery, an expected average of 12 hours
  Number of attempts to place the tracheal tube via fiberoptic bronchoscopy through supraglottic device will be limited to 3

CONTACTS AND LOCATIONS:
Overall Officials: Narasimhan Jagannathan, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago / Stanley Manne Research Institute
Locations (1):
- Anne & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Timmermann A. Supraglottic airways in difficult airway management: successes, failures, use and misuse. Anaesthesia. 2011 Dec;66 Suppl 2:45-56. doi: 10.1111/j.1365-2044.2011.06934.x. PMID 22074079
- [Background] Sohn LE, Jagannathan N, Sequera-Ramos L, Sawardekar A, Schaldenbrand K, De Oliveira GS. A randomised comparison of free-handed vs air-Q assisted fibreoptic-guided tracheal intubation in children < 2 years of age. Anaesthesia. 2014 Jul;69(7):723-8. doi: 10.1111/anae.12667. Epub 2014 May 2. PMID 24797607
- [Background] Mathis MR, Haydar B, Taylor EL, Morris M, Malviya SV, Christensen RE, Ramachandran SK, Kheterpal S. Failure of the Laryngeal Mask Airway Unique and Classic in the pediatric surgical patient: a study of clinical predictors and outcomes. Anesthesiology. 2013 Dec;119(6):1284-95. doi: 10.1097/ALN.0000000000000015. PMID 24126262
- [Background] Abukawa Y, Hiroki K, Ozaki M. Initial experience of the i-gel supraglottic airway by the residents in pediatric patients. J Anesth. 2012 Jun;26(3):357-61. doi: 10.1007/s00540-011-1322-1. Epub 2012 Feb 7. PMID 22310833
- [Background] Foucher-Lezla A, Lehousse T, Monrigal JP, Granry JC, Beydon L. Fibreoptic assessment of laryngeal positioning of the paediatric supraglottic airway device I-Gel. Eur J Anaesthesiol. 2013 Jul;30(7):441-2. doi: 10.1097/EJA.0b013e32835f9969. No abstract available. PMID 23571478
- [Background] Hughes C, Place K, Berg S, Mason D. A clinical evaluation of the I-gel supraglottic airway device in children. Paediatr Anaesth. 2012 Aug;22(8):765-71. doi: 10.1111/j.1460-9592.2012.03893.x. Epub 2012 Jun 1. PMID 22672411
- [Background] Jagannathan N, Sommers K, Sohn LE, Sawardekar A, Shah RD, Mukherji II, Miller S, Voronov P, Seraphin S. A randomized equivalence trial comparing the i-gel and laryngeal mask airway Supreme in children. Paediatr Anaesth. 2013 Feb;23(2):127-33. doi: 10.1111/pan.12078. Epub 2012 Nov 27. PMID 23189931
- [Background] Emmerich M, Tiesmeier J. The I-gel supraglottic airway: a useful tool in case of difficult fiberoptic intubation. Minerva Anestesiol. 2012 Oct;78(10):1169-70. No abstract available. PMID 23059523
- [Background] Kim YL, Seo DM, Shim KS, Kim EJ, Lee JH, Lee SG, Ban JS. Successful tracheal intubation using fiberoptic bronchoscope via an I-gel supraglottic airway in a pediatric patient with Goldenhar syndrome -A case report-. Korean J Anesthesiol. 2013 Jul;65(1):61-5. doi: 10.4097/kjae.2013.65.1.61. Epub 2013 Jul 19. PMID 23904941
- [Background] Kim MS, Oh JT, Min JY, Lee KH, Lee JR. A randomised comparison of the i-gel and the Laryngeal Mask Airway Classic in infants. Anaesthesia. 2014 Apr;69(4):362-7. doi: 10.1111/anae.12592. PMID 24641642
- [Background] Jagannathan N, Sohn LE, Sawardekar A, Gordon J, Shah RD, Mukherji II, Roth AG, Suresh S. A randomized trial comparing the Ambu (R) Aura-i with the air-Q intubating laryngeal airway as conduits for tracheal intubation in children. Paediatr Anaesth. 2012 Dec;22(12):1197-204. doi: 10.1111/pan.12024. Epub 2012 Sep 13. PMID 22971118
- [Background] Park C, Bahk JH, Ahn WS, Do SH, Lee KH. The laryngeal mask airway in infants and children. Can J Anaesth. 2001 Apr;48(4):413-7. doi: 10.1007/BF03014975. PMID 11339788
- [Derived] Jagannathan N, Sohn L, Ramsey M, Huang A, Sawardekar A, Sequera-Ramos L, Kromrey L, De Oliveira GS. A randomized comparison between the i-gel and the air-Q supraglottic airways when used by anesthesiology trainees as conduits for tracheal intubation in children. Can J Anaesth. 2015 Jun;62(6):587-94. doi: 10.1007/s12630-014-0304-9. Epub 2014 Dec 24. PMID 25537736